CLINICAL TRIAL: NCT06591364
Title: Prevalence and Predictive Factors of Difficult Biliary Cannulation: a Multicenter Study
Brief Title: Prevalence and Predictive Factors of Difficult Biliary Cannulation
Acronym: PRECABIDO
Status: Not yet recruiting | Type: Observational
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Clinical Professor, University of La Laguna
Other Study IDs: PRECABIDO
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Difficult Biliary Cannulation
Keywords: ERCP; Endoscopic retrograde cholangiopancreatography; Difficult biliary cannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main purpose of the study is to evaluate the prevalence of difficult biliary cannulation using endoscopic retrograde cholangiopancreatography (ERCP) according to the criteria defined by the European Society of Gastrointestinal Endoscopy (ESGE) and the American Society for Gastrointestinal Endoscopy (ASGE), as well as the predictive factors for this event in a prospective, multicenter study. Consecutive patients undergoing ERCP will be included in the study

We will also assess:

Evaluate the failure of biliary cannulation in our setting. Evaluate predictive factors for difficult cannulation and cannulation failure using ESGE criteria.

Design an "a priori" predictive model for difficult cannulation and cannulation failure.

Cost study: record of materials used.

DETAILED DESCRIPTION:
All consecutive patients who meet the inclusion criteria and none of the exclusion criteria will be offered participation in the study. They will be informed by one of the investigators from each center and will sign an informed consent form. A data collection sheet will be completed to record demographic data, the indication for the procedure, and technical variables.

The procedures will be performed by endoscopists with at least 200 ERCPs and more than 5 years of experience. All patients, except in cases of allergy, will receive 1 suppository of indomethacin or diclofenac before the procedure. In cases of allergy, pre-procedure hydration with Ringer's lactate will be administered if there is no contraindication (consider the protocol proposed by the ESGE: 3 mL/kg/hour during ERCP, 20 mL/kg as a bolus after ERCP, and 3 mL/kg/hour for 8 hours post-ERCP). The use of a pancreatic stent should be considered when indicated.

After the procedure, patients will remain hospitalized for at least 24 hours in the hospital. The patient's medical record will be reviewed 7 days after the procedure to check for any adverse effects, and a follow-up phone call will be made to detect any adverse effects.

Initially, a pilot study will be conducted with 600 patients, assessing based on the results-that is, the percentage of patients with difficult cannulation and the number of independent variables associated in the multiple logistic regression-the need to include a larger number of patients. For each variable included in the multiple logistic regression analysis, 8 to 10 cases of patients with difficult cannulation would be required.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed informed consent
* Patients indicated for ERCP

Exclusion Criteria:

* INR > 1.5
* Platelets < 50,000/mm³
* Patients with a prior endoscopic sphincterotomy
* Papilla of Vater not accessible via duodenoscope (gastric or duodenal stenosis due to neoplasm) or gastric surgery (Billroth II, Roux-en-Y)
* Known pancreas divisum
* Indication due to pancreatic duct pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive patients with an indication of a endoscopic retrograde cholangiopancreatography meeting inclusion and exclusion criteria will be included
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Difficult biliary cannulation | 1 year
  (> 5 minutes duration until cannulation, > 5 cannulation attempts, > 1 passage of the guidewire into the main pancreatic duct

SECONDARY OUTCOMES:
Failure of biliary cannulation | 1 year
  Not possibility of biliary cannulation during the procedure
Predictive factors for difficult cannulation and cannulation failure | 1 year
  Factors independently associated with difficult cannulation and cannulation failure
Designing an "a priori" predictive model for difficult cannulation and cannulation failure | 1 year
  Considering the factors independently associated with difficult cannulation and cannulation failure
To carry out a cost study | 1 year
  considering direct costs of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno García, MD, PhD, Principal Investigator — University Hospital of the Canary Islands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baron TH, Petersen BT, Mergener K, Chak A, Cohen J, Deal SE, Hoffinan B, Jacobson BC, Petrini JL, Safdi MA, Faigel DO, Pike IM; ASGE/ACG Taskforce on Quality in Endoscopy. Quality indicators for endoscopic retrograde cholangiopancreatography. Am J Gastroenterol. 2006 Apr;101(4):892-7. doi: 10.1111/j.1572-0241.2006.00675.x. No abstract available. PMID 16635233
- [Background] Caceres-Escobar D, Munoz-Velandia OM, Vargas-Rubio R. FACTORS ASSOCIATED WITH DIFFICULT BILIARY CANNULATION IN A TRAINING CENTER FOR ENDOSCOPIC INTERVENTION OF THE BILIARY TRACT. Arq Gastroenterol. 2022 Jan-Mar;59(1):29-34. doi: 10.1590/S0004-2803.202200001-06. PMID 35442332
- [Background] Dalal A, Gandhi C, Patil G, Kamat N, Vora S, Maydeo A. Safety and efficacy of different techniques in difficult biliary cannulation at endoscopic retrograde cholangiopancreatography. Hosp Pract (1995). 2022 Feb;50(1):61-67. doi: 10.1080/21548331.2022.2029451. Epub 2022 Jan 20. PMID 35025705
- [Background] Saito H, Kadono Y, Shono T, Kamikawa K, Urata A, Nasu J, Imamura H, Matsushita I, Kakuma T, Tada S. Factors Predicting Difficult Biliary Cannulation during Endoscopic Retrograde Cholangiopancreatography for Common Bile Duct Stones. Clin Endosc. 2022 Mar;55(2):263-269. doi: 10.5946/ce.2021.153. Epub 2021 Nov 12. PMID 34763384